CLINICAL TRIAL: NCT06041607
Title: Shared Meditation Involving People With Cancer, Carers and Third Parties: Any Added Value Compared With Meditation Conducted With Patients? IMPLIC 2, a Randomised Study
Brief Title: Shared Meditation Involving People With Cancer, Carers and Third Parties
Acronym: IMPLIC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A01373-42
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Patients With Cancer
Keywords: meditation; carer
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared meditation (Experimental): Shared" meditation: mixed groups of patients, carers and third parties
  Interventions: Behavioral: Shared meditation
- Meditation "patients" (Active Comparator): groups of patients only
  Interventions: Behavioral: Meditation with patients oly

INTERVENTIONS:
Behavioral: Shared meditation — Meditation sessions between patients, carers and third parties
  * 12 weekly 2-hour sessions,
  * 2 half-day 3-hour retreats after the 9th session and at the end of the programme
  * 3 monthly follow-up sessions (2h) in remote format (videoconference)
  Arms: Shared meditation
Behavioral: Meditation with patients oly — Meditation sessions between patients only
  * 12 weekly 2-hour sessions,
  * 2 half-day 3-hour retreats after the 9th session and at the end of the programme
  * 3 monthly follow-up sessions (2h) in remote format (videoconference)
  Arms: Meditation "patients"

SUMMARY:
Although the benefits of meditation are increasingly well documented, few hospitals offer this integrative approach in their supportive cancer care. Meditation is sometimes provided, but its potential benefits remain insufficiently evaluated.

This project is based on the hypothesis that there could be a benefit in meditating together.

DETAILED DESCRIPTION:
The main aims of this randomised study are to improve well-being, strengthen links between carers, patients and third parties and raise awareness of the importance of living together better by offering meditation as a shared activity. The expected benefits of meditation therefore primarily concern the relief of psychological suffering. Promoting better understanding between carers and patients, and looking at oneself and others in a different way are experiences that aim to encourage exchanges and interactions between populations. For cancer patients (the target population), pain and other symptoms associated with the disease and its treatment will be better managed.

The pain experienced by carers, which is essentially linked to professional overwork and contact with illness, will be considered and managed through meditation, resulting in benefits for carers and their way of interacting with their patients.

The expected collective benefit is to develop and better live together our interdependence and humanity, by recognising suffering as a shared characteristic, despite our specific problems (as patients, carers or third parties).

The overall aim is to alleviate suffering, which is an integral part of the human experience, by cultivating our common humanity.

ELIGIBILITY:
Inclusion Criteria:

Criteria for all participants (patients, carers and third parties)

* Participant with no current or previous experience of regular or intensive meditation or comparable practice. Practice is considered regular and/or intensive if :
* it occurs more than one day a week for more than 6 consecutive months over the last 10 years,
* and/or more than 5 consecutive days of intensive practice (course or retreat) in the last 10 years,
* and/or more than 25 consecutive days of retreat (cumulative) in the last 10 years.

Patient-specific criteria (target population) - Cancer patients (regardless of location)

Specific criteria for carers

- All medical and/or paramedical care staff at the Centre François Baclesse in contact with patients (doctors, nurses, nursing assistants, radiotherapy technicians, etc.)

Specific criteria for third parties- Any volunteer not belonging to the two categories above

Exclusion Criteria:

* Participants with significant vulnerability factors such as alcohol or drug dependence, severe depression, severe social anxiety, recent bereavement, etc.)
* Participant unable to undergo trial monitoring for geographical, social or psychopathological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
To assess the possible added value for patients (target population) of a meditation programme shared between patients, carers and third parties, compared with the same meditation programme conducted solely for patients. | measured at the end of the meditation programme (after the 12 weekly sessions) compared with the measurement at inclusion
  Changes in self-efficacy scores according to the Generalized Self Efficacy Scale [min 10; max 40]

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prevost V, Tran T, Leconte A, Lequesne J, Fernette M, Segura C, Chevigne S, Gouriot M, Clarisse B. A randomised study to evaluate the potential added value of shared meditation involving people with cancer, health professionals and third persons compared to meditation conducted with patients only: design of the Implic-2 protocol. BMC Cancer. 2024 Sep 4;24(1):1097. doi: 10.1186/s12885-024-12521-1. PMID 39232668